CLINICAL TRIAL: NCT03999710
Title: Durvalumab With Thoracic Radiation Therapy Without Chemotherapy for Locally Advanced Non-Small Cell Lung Cancer (DART)
Brief Title: Determining Whether Durvalumab in Combination With Radiation Therapy Can Prevent the Progression of Non-Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-218
Record Dates: First submitted 2019-06-25; First posted 2019-06-27 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Non Small Cell Lung Cancer; Lung Cancer; Nsclc; NSCLC Stage II; NSCLC, Stage III
Keywords: Lung Cancer; Non Small Cell Lung Cancer; Radiation therapy; durvalumab; 19-218; Memorial Sloan Kettering Cancer Center; newly diagnosed; recurrent
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Recurrence | interventions — Radiotherapy; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Non-Small Cell Lung Cancer (Experimental): All participants have locally-advanced non-small cell lung cancer, Stage II-III. Treatment will consist of durvalumab administered concurrently with thoracic radiation consisting of 60 Gy in 30 fractions. Patients will be monitored weekly during on-treatment visits. Durvalumab will then be continued up to 1 year as maintenance or until disease progression or unacceptable toxicity. Optional Research MRIs (Does not apply to the Alliance Sites. Research MRIs will only be done at MSKCC)
  Interventions: Radiation: Radiation Therapy; Drug: Durvalumab

INTERVENTIONS:
Radiation: Radiation Therapy — Treatment will consist of 60 Gy in 30 fractions to fields encompassing gross tumor and lymph nodes.
Drug: Durvalumab — A dose of 1500mg (for patients >30kg in weight) will be administered using an IV bag containing 0.9% (w/v) saline or 5% (w/v) dextrose, with a final durvalumab concentration ranging from 1 to 15 mg/mL, and delivered through an IV administration set with a 0.2- or 0.22- μm filter.

SUMMARY:
The purpose of this study is to see if Durvalumab and radiation therapy can delay the worsening of disease in patients with non-small cell lung cancer normally treated with sequential chemotherapy followed by radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
* Patient age >/= 18 at time of consent
* Newly diagnosed or recurrent Locally-advanced NSCLC (stage II-III) amenable for treatment with concurrent definitive radiation and durvalumab
* Ineligible for resection and concurrent CRT as determined by one of the following reasons: Medically inoperable, surgically unresectable (including N3 nodal disease), medically unfit or unsafe for chemotherapy, or other reason deemed appropriate by the investigator and approved by PI.

Note: The reason a patient is deemed ineligible for concurrent CRT must be documented (i.e. hearing impairment, neuropathy, renal dysfunction, symptomatic/advanced underlying medical comorbidities, etc.)

* Histological and/or cytological confirmation of NSCLC (both squamous and adenocarcinoma) as per standard of care biopsy; no additional research protocol-specific biopsy is needed.
* ECOG/WHO PS 0-2
* Candidates for definitive RT to 60 Gy in 30 fractions
* Body weight > 30kg
* Adequate normal organ and marrow function as defined below:

  * Hemoglobin >/= 9.0 g/dL
  * Absolute neutrophil count (ANC) 1.5 x (>/= 1500 per mm3)
  * Platelet count >/= 75 x 10^9/L (>/= 75,000 per mm3)
  * Serum bilirubin </= 1.5 x institutional upper limit of normal (ULN). This will not apply to patients with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
  * AST (SGOT)/ALT (SGPT) </= 2.5 x institutional upper limit of normal
  * Measured creatinine clearance (CL) >15mL/min or Calculated creatinine CL>15 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance.

Males:

Creatinine CL (mL/min) = [Weight (kg) x (140 - Age)] / [72 x serum creatinine(mg/dL)]

Females:

Creatinine CL (mL/min) = [Weight (kg) x (140 - Age)] / [72 x serum creatinine(mg/dL)] x 0.85

* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply.

  * Women >/= 50 years of age would be considered would be considered post-menopausal if they have been amenorrheic for 12 months following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy)
  * Women >/= 50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses > 1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy)
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Must have a life expectancy of at least 12 weeks

Exclusion Criteria:

* Participants in another clinical study with an investigational product during the last 4 weeks
* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
* Previous thoracic radiation precluding definitive RT
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], acute diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

  1. Patients with vitiligo or alopecia
  2. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  3. Any chronic skin condition that does not require systemic therapy
  4. Patients without active disease in the last 5 years may be included but only after consultation with the study physician
  5. Patients with celiac disease controlled by diet alone
* Any unresolved toxicity NCI CTCAE Grade >/=2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

  1. Patients with Grade >/= neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician
  2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.
* Prior/Current Therapies

  1. Treatment with a monoclonal antibody within 4 weeks prior to study Day 1 or has not recovered (i.e., >/= Grade 1 at baseline) from adverse events due to agents administered > 4 weeks earlier (intraocular bevacizumab is acceptable)
  2. Prior chemotherapy or targeted small molecule therapy, within 3 weeks prior to study Day 1 or has not recovered (i.e., >/= Grade 1 at baseline) from adverse events due to a previously administered agents (excluding Grade 2 peripheral neuropathy)
  3. Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLAA-4) antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
  4. Current or prior use of immunosuppressive medication within 7 days before the first dose of durvalumab. The following are exceptions to this criterion:

  i. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection) ii. Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent iii. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication) e. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.

  f. Prior chemotherapy for this diagnosis of lung cancer.
* Major surgical procedure (as defined by the investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
* History of allogenic organ transplantation
* Severe concurrent illness:

  1. Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trials.
  2. Known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
  3. Active known infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice) or hepatitis B (known positive HBV surface antigen (HBsAg) result). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA. Testing for Hepatitis C and HIV is not required unless clinically indicated.
  4. Evidence of interstitial lung disease or active, non-infectious pneumonitis
  5. Clinically significant (i.e., active) cardiovascular disease: symptomatic cerebral vascular accident/stroke (< 6 months prior to enrollment) with out neurological recovery, unstable angina, congestive heart failure (≥ New York Heart Association Classification Class III), or serious cardiac arrhythmia uncontrolled with current medication.
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ a highly effective birth control from screening to 90 days after the last dose of durvalumab monotherapy

  a. Highly effective methods of contraception, defined as one that results in a low failure rate (ie, less than 1% per year) when used consistently and correctly are described in Table 1. Note that some contraception methods are not considered highly effective (e.g. male or female condom with or without spermicide; female cap, diaphragm, or sponge with or without spermicide; non-copper containing intrauterine device; progestogen-only oral hormonal contraceptive pills where inhibition of ovulation is not the primary mode of action [excluding Cerazette/desogestrel which is considered highly effective]; and triphasic combined oral contraceptive pills).

  i. Barrier/Intrauterine Methods: Copper T intrauterine device; Levonorgestrel-releasing intrauterine system (e.g., Mirena) ii. Hormonal Methods: Implants - Etonogestrel-releasing implants (e.g. Implanon or Norplant); Intravaginal - Ethinylestradiol/etonogestrel-releasing intravaginal devices (e.g., NuvaRing); Injection - Medroxyprogesterone (e.g., Depo-Provera); Combined Pill - normal and low dose combined oral contraceptive pill; Patch - Norelgestromin/ethinylestradiol-releasing transdermal system (e.g., Ortho Evra); Minipills: Progesterone based oral contraceptive pill using desogestrel (Cerazette is currently the only highly effective progesterone-based)
* Live vaccination with 4 weeks prior to the first dose of durvalumab and while on trial is prohibited except for administration of inactivated vaccines
* Connective tissue disorders involving the lung(s) and/or esophagus requiring active treatment or idiopathic pulmonary fibrosis
* Known actionable EGFR or ALK mutation
* Known contraindications to radiotherapy
* Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
2-year PFS rate | 2 years
  Demonstrate an improvement in 2-year PFS rate compared to historical results.

CONTACTS AND LOCATIONS:
Overall Officials: Narek Shaverdian, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - Baptist Alliance Miami Cancer Institute, Miami, Florida
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Lehigh Valley Health Network, Allentown, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org